CLINICAL TRIAL: NCT00001625
Title: Methods for Assessing Insulin Sensitivity In Vivo
Brief Title: Methods for Measuring Insulin Sensitivity
Status: Completed | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: Office of Dietary Supplements (ODS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970105; 97-AT-0105
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-04-11

CONDITIONS: Obesity; Hypertension; Diabetes-Mellitus, Non-Insulin Dependent
Keywords: Insulin Resistance; Obesity; Hypertension; Diabetes; Mathematical Modeling; Normal Volunteer
MeSH Terms: conditions — Obesity; Hypertension; Diabetes Mellitus, Type 2; Insulin Resistance; Diabetes Mellitus

SUMMARY:
Patients with high blood pressure, diabetes, and who are overweight are known to have defects in the way their body responds to insulin. The purpose of this study is to develop better methods for measuring the way body tissue responds to insulin and sugar (glucose).

Researchers are planning to study four groups of patients.

1. Normal volunteers
2. Patients who have mild to moderate high blood pressure
3. Patients who are overweight
4. Patients who have mild to moderate diabetes controlled with oral medication

In this study patients and volunteers will undergo two separate tests designed to determine how well insulin is working in the body. The first test is called a glucose clamp test. Patients will have two needles placed in the veins of their arms. One needle will be used to take blood samples, the other needle will be used to inject doses of sugar (glucose) and insulin.

The second test is called the frequently sample intravenous glucose tolerance test. In this test patients will have sugar (glucose) injected into their veins followed by a slow injected dose (infusion) of insulin. Researchers will periodically take blood samples during the test.

Patients participating in the study will not directly benefit from it. However, the information gained from this study may be useful for improving the diagnosis and therapy of diseases such as diabetes, obesity, and high blood pressure (hypertension).

DETAILED DESCRIPTION:
We hypothesize that the majority of the information needed to accurately estimate insulin sensitivity is contained in the fasting insulin and glucose levels as well as the insulin and glucose levels obtained shortly after an intravenous glucose load. We propose to test this hypothesis by performing both hyperinsulinemic euglycemic glucose clamps as well as intravenous glucose tolerance tests on normal volunteers and groups of patients with diabetes, hypertension, or obesity (diseases known to be associated with insulin resistance). Data from these studies will be used obtain estimates of insulin sensitivity by the glucose clamp method, minimal model method, and a novel analysis that utilizes only fasting and peak levels of glucose and insulin. We hope to devise a simpler method for determining insulin sensitivity in vivo that is suitable for testing large populations. This method will require only a few blood samples, take less than one hour to perform, and correlate with glucose clamp estimates at least as well as the minimal model method.

ELIGIBILITY:
* INCLUSION CRITERIA:

Normal Volunteers:

Adults between the ages of 21 and 55 in good general health with no significant underlying illnesses, on no medication, and a normal body mass index (20-26 kg/m(2)).

Obese Subjects:

Adults between the ages of 21 and 55 in good general health with no significant underlying illnesses, on no medication, and a body mass index between 30 and 35 kg/m(2).

Hypertensive Subjects:

Adults between the ages of 21 and 55 in good general health except for mild to moderate hypertension (blood pressure between 140/95 and 170/109 off medication), on no medication except for antihypertensive agents.

Subjects will be taken off all antihypertensive drugs for at least one week prior to study. If a subjects blood pressure exceeds 180/110 on three determinations over a period of at least 15 minutes, the subject will be withdrawn from the study and appropriate antihypertensive therapy resumed.

Diabetic Subjects:

Adults between the ages of 21 and 65 in good general health except for non-insulin dependent diabetes mellitus controlled with oral hypoglycemic agents. Subjects on no other medications. If fasting blood glucose exceeds 300 mg/dl, the subject will be withdrawn from the study and appropriate therapy resumed.

EXCLUSION CRITERIA:

Pregnancy, liver disease, pulmonary disease, end-organ damage such as renal insufficiency, coronary artery disease, heart failure, peripheral vascular disease, proliferative retinopathy, diabetic neuropathy, or HIV infection.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480
Dates: Start 1997-04-03; Study Completion 2007-04-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Quon MJ, Cochran C, Taylor SI, Eastman RC. Non-insulin-mediated glucose disappearance in subjects with IDDM. Discordance between experimental results and minimal model analysis. Diabetes. 1994 Jul;43(7):890-6. doi: 10.2337/diab.43.7.890. PMID 8013753